CLINICAL TRIAL: NCT03574818
Title: A Feasibility and Biomarker Study to Evaluate Necitumumab in the Neoadjuvant Setting With Gemcitabine and Cisplatin in Surgically Resectable Squamous Lung Cancer
Brief Title: Necitumumab in the Neoadjuvant Setting With Gemcitabine in Surgically Resectable - 14X-US-I001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Montefiore Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Balazs Halmos, Director of Thoracic Oncology / Assistant Professor of Medicine, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-8108
Record Dates: First submitted 2018-04-24; First posted 2018-07-02 (Actual); Results first posted 2020-02-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Neoadjuvant Chemotherapy; NSCLC; nacitumumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Feasibility and Biomaker Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Chemotherapy and Necitumumab Regimen Gemcitabine 1250mg/m2 IV over 30 minutes, days 1 and 8 following necitumumab, Cisplatin 75mg/m2 IV over 60 minutes, day 1, immediately following gemcitabine,each cycle is 3 weeks (21 days).
  Necitumumab 800mg absolute dose IV over a minimum of 60 minutes, days 1 and 8 prior to chemotherapy regimen Each cycle is 3 weeks (21 days).
  The regimen will be given for a total of 3 cycles.
  The regimen will be given for a total of 3 cycles.
  Interventions: Drug: Necitumumab-Gemcitabine-Cisplatin; Diagnostic Test: Evaluation to determine if patient is a candidate to proceeed with surgical resection or not

INTERVENTIONS:
Drug: Necitumumab-Gemcitabine-Cisplatin — * Gemcitabine 1250mg/m2 IV on D1, D8
  * Cisplatin 75mg / m2 IV on D1
  * Necitumumab 800mg IV on D1, D8 (peripheral blood for effector cells and cytokine measurements prior to each cycle) Repeat cycle every 21 days up to 3 cycles.
  Other Names: PORTRAZZA™ - GEMZAR™ - PLATINOL™
Diagnostic Test: Evaluation to determine if patient is a candidate to proceeed with surgical resection or not — Patients will be evaluated with repeat imaging studies (PET/CT or CT Chest, Abdomen, Pelvis) and will be re-evaluated for surgical resection. Patients who had progressive disease or are NOT a surgical candidate will come off the study and will be treated according to standard therapies. All patients will be followed up for 2-year disease-free survival and overall survival

SUMMARY:
This will be a single-arm study to primarily evaluate the feasibility of administering necitumumab added to gemcitabine and cisplatin as neoadjuvant treatment in treatment-naïve patients with stage IB (tumor size >4cm), II or IIIA squamous NSCLC. Feasibility will be assessed by the proportion of patients able to proceed to surgery after administering necitumumab in the neoadjuvant setting. These patients would otherwise be offered standard adjuvant chemotherapy (without necitumumab) for squamous cell lung cancer. Determination of surgical resectability will be reviewed at a multidisciplinary thoracic tumor board, attended by surgical oncology, medical oncology, radiation oncology, radiology, and pathology.

DETAILED DESCRIPTION:
The goal of this study is to explore whether it is possible to add a drug called necitumumab to standard treatment for patients with squamous cell lung cancer that can be surgically removed. This study is important because it will determine whether there is added benefit to giving necitumumab with chemotherapy before surgery. It is currently already known that chemotherapy given before or after surgery has better outcomes compared to only receiving surgery. Results from this study may help to develop more effective treatments for patients with squamous cell lung cancer.

The U.S. Food and Drug Administration (FDA) has approved necitumumab in combination with chemotherapy drugs called gemcitabine and cisplatin to treat stage IV or metastatic squamous cell lung cancer, but the FDA has not approved necitumumab to treat squamous cell lung cancer that can be surgically removed.

Analyzing the tumor cells from many cases of squamous cell lung cancer has shown that this cancer often has a special protein called EGFR. Necitumumab is a drug that targets EGFR.

Results from a recent medical study showed that patients with stage IV or metastatic squamous cell lung cancer who received necitumumab with gemcitabine and cisplatin showed a small, but significant, improvement in survival. We believe trying to gather more information about the way necitumumab interacts with cancer cells will help to learn how to use necitumumab more effectively.

This study will allow to see the effects of treating an earlier stage of squamous cell lung cancer using necitumumab with gemcitabine and cisplatin. It will also allow us to better analyze tumor cells after they have been treated with necitumumab and chemotherapy that are obtained after surgical resection. Other blood samples that will be drawn during the treatment will also allow to see the effect of necitumumab on both the body and the tumor cells and to observe any side effects that may result from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell non-small cell lung cancer with any of the following stage groupings: IB with tumor size >4cm, II or potentially resectable IIIA.
* Patients who have been evaluated by thoracic surgery and eligible for resection.
* Patients must have adequate fresh frozen paraffin embedded (FFPE) tumor tissue available to perform pre-treatment biomarker testing.
* No prior systemic treatment for squamous cell non-small cell lung cancer.
* Age ≥18 years.
* ECOG performance status 0-1 (Karnofsky ≥70%, see Appendix A).
* Patients must have hematologic function as defined by:

  * absolute neutrophil count ≥1.5 x 109/L
  * hemoglobin ≥9.0 g/dL
  * platelets ≥100 x 109/L
* Patients must have organ function as defined below:

  * bilirubin ≤1.5 × the upper limit of normal (ULN), alkaline phosphatase (ALP), alanine aminotransferase (ALT) and asparate transaminase (AST) ≤3.0 times ULN. For patients with hepatic metastases, ALT and AST equaling ≤5.0 times ULN are acceptable.
  * If a patient experiences elevated ALT >5 × ULN and elevated total bilirubin >2 × ULN, clinical and laboratory monitoring should be initiated by the investigator. For patients entering the study with ALT >3 × ULN, monitoring should be triggered at ALT >2 × baseline.
  * calculated creatinine clearance >50mL/min (per the Cockcroft-Gault formula).
  * serum albumin ≥2.5 g/dL
* Patients may be on a stable regimen of therapeutic anticoagulation or may be receiving prophylactic anticoagulation of venous access devices.
* The patient is a woman of child-bearing potential who tests negative for pregnancy within 14 days prior to receiving first dose of study medication based on serum pregnancy test and agrees to use 2 methods of birth control or abstain from heterosexual activity during the study and for 6 months following the last dose of the study drug(s) or country requirements, whichever is longer or be of non-child bearing potential.
* Non-childbearing potential is defined as (by other than medical reasons):

  * ≥45 years of age and has not had menses for greater than 2 years,
  * amenorrheic for < 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation, or
  * post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 6 months after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.
* The patient is willing to comply with protocol schedules and testing. -
* Exclusion Criteria: Patients with histologically or cytologically confirmed non-squamous cell, small cell or mixed histology lung carcinoma.
* Patients with stage IIIB or stage IV disease.
* Prior history of other malignancy, provided that he/she has been free of disease for ≥3 years, with the exception of in-situ carcinoma of the cervix or completely resected basal cell carcinoma of the skin.
* Patients who are receiving any other investigational agents.
* The patient has a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab, or any other contraindication to one of the administered treatments.
* History or evidence of current clinically relevant coronary artery disease ≥ Grade III by the Canadian Cardiovascular Society Angina Grading Scale or uncontrolled congestive heart failure of current > Class III as defined by the New York Heart Association.
* The patient has experienced myocardial infarction within 6 months prior to study enrollment.
* The patient has any ongoing or active infection, including active tuberculosis or known infection with the human immunodeficiency virus.
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination.
* The patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.
* History of arterial or venous thromboembolism within 3 months prior to study enrollment. Patients with a history of venous thromboembolism beyond 3 months prior to study enrollment can be enrolled if they are appropriately treated with low molecular weight heparin.
* The patient has any NCI-CTCAE Version 4.0 Grade ≥2 peripheral neuropathy.
* The patient has any other serious uncontrolled medical disorders or psychological conditions that would, in the opinion of the investigator, limit the patient's ability to complete the study or sign an informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: one patient was enrolled in May 2018, study was terminated in September 2019 due to poor accrual
Groups:
- Arm 1: Chemotherapy and Necitumumab Regimen Gemcitabine 1250mg/m2 IV over 30 minutes, days 1 and 8 following necitumumab, Cisplatin 75mg/m2 IV over 60 minutes, day 1, immediately following gemcitabine,each cycle is 3 weeks (21 days).
  Necitumumab 800mg absolute dose IV over a minimum of 60 minutes, days 1 and 8 prior to chemotherapy regimen Each cycle is 3 weeks (21 days).
  The regimen will be given for a total of 3 cycles.
  The regimen will be given for a total of 3 cycles.
  Necitumumab-Gemcitabine-Cisplatin: / Gemcitabine 1250mg/m2 IV on D1, D8
  * Cisplatin 75mg / m2 IV on D1
  * Necitumumab 800mg IV on D1, D8 (peripheral blood for effector cells and cytokine measurements prior to each cycle) Repeat cycle every 21 days up to 3 cycles.
Period: Overall Study
Arm/Group | Arm 1
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Surgically Resectable
Description: Patients able to proceed to surgery after administering necitumumab in the neoadjuvant setting with gemcitabine and cisplatin in surgically resectable patients with stage IB with tumor size >4cm, II and potentially resectable IIIA squamous cell lung cancer.
Time Frame: up to 63 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: neoadjuvant treatment period - up to 63 days
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1 rash
mucositis (Gastrointestinal disorders) | 1 (1) — grade 1 mucositis
hypomagnesemia (Investigations) | 1 (1) — grade 2 hypomagnesemia
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1 cough
neutropenia (Blood and lymphatic system disorders) | 1 (1) — grade 3 neutropenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03574818/Prot_SAP_ICF_000.pdf